CLINICAL TRIAL: NCT02410499
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled, Proof of Concept, Phase 2 Study to Evaluate the Efficacy and Safety of Weekly Subcutaneous MLN1202, in Improving Diabetic Nephropathy in Subjects With Macroalbuminuria
Brief Title: Efficacy and Safety of Weekly Subcutaneous MLN1202 in Improving Diabetic Nephropathy in Participants With Macroalbuminuria
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN1202-2005; 2014-005142-21 (EudraCT Number); U1111-1168-1426 (Registry Identifier: WHO Universal Trial Number)
Record Dates: First submitted 2015-04-02; First posted 2015-04-07 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Diabetic Nephropathy
Keywords: Drug therapy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — plozalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): MLN1202 placebo-matching solution, subcutaneous injection (SC), once, on Day 1 (loading dose), followed by MLN1202 placebo-matching solution, SC, once, weekly, on Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: MLN1202 Placebo
- MLN1202 75 mg (Experimental): MLN1202 450 mg, solution, SC injection, once, on Day 1 (loading dose), followed by MLN1202 75 mg, solution, SC, once, weekly, on Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: MLN1202
- MLN1202 105 mg (Experimental): MLN1202 450 mg, solution, SC injection, once, on Day 1 (loading dose), followed by MLN1202 105 mg, solution, SC, once, weekly, on Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: MLN1202
- MLN1202 150 mg (Experimental): MLN1202 450 mg, solution, SC injection, once, on Day 1 (loading dose), followed by MLN1202 150 mg, solution, SC, once, weekly, on Days 8, 15, 22, 29, 36, 43, 50, 57, 64, 71, and 78.
  Interventions: Drug: MLN1202

INTERVENTIONS:
Drug: MLN1202 Placebo — MLN1202 placebo-matching solution for SC injection
  Arms: Placebo
Drug: MLN1202 — MLN1202 solution for SC injection
  Arms: MLN1202 105 mg; MLN1202 150 mg; MLN1202 75 mg

SUMMARY:
The purpose of this study is to characterize the effects of 85 days treatment with MLN1202 on urinary albumin-to-creatinine ratio (UACR) in participants with type 2 diabetes, advanced kidney disease/diabetic nephropathy (DN) and macro-albuminuria (UACR>300 mg/g) based on average of 3 consecutive first morning voids sample collection.

DETAILED DESCRIPTION:
The drug being tested in this study is called MLN1202. MLN1202 is being tested to treat people who have diabetes with macroalbuminuria. This study will look at the urinary albumin-to-creatinine ratio in people who take MLN1202.

The study will enroll approximately 156 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the four treatment groups-which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* MLN1202 75 mg subcutaneous (SC) injection
* MLN1202 105 mg SC injection
* MLN1202 150 mg SC injection
* Placebo matching MLN1202 SC injection (dummy inactive solution) - this is a solution that looks like the study drug but has no active ingredient

All participants will receive a loading dose of placebo or MLN1202 on Day 1 followed by once-weekly injections of the study medication they were randomized to receive.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is 5 months. Participants will make multiple visits to the clinic, plus a final visit 5 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of giving informed consent to enter the trial, including understanding and complying with protocol requirements.
2. The participant or, when applicable, (eg, where the subject is capable of giving verbal informed consent to enter the trial but cannot physically sign a written, informed consent form), the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
3. At the time of Screening the participant is male or female and aged 18-90 years inclusive at first dose of study medication.
4. Was previously diagnosed with type 2 diabetes mellitus per American Diabetes Association criteria.
5. Has an estimated glomerular filtration rate (eGFR) based on serum creatinine (eGFR, determined by Modification of Diet in Renal Disease [MDRD] equation) of 25-59 mL/min/1.73 m(2) at Screening.
6. Has been on a stable dose of angiotensin-converting enzyme (ACE) inhibitor or angiotensin II receptor blocker (ARB) for 8 weeks prior to Screening.
7. Has residual albuminuria despite stable treatment with an ACE inhibitor or an ARB for at least 8 weeks prior to Screening (albumin:creatinine ratio [ACR] of > 300 mg/g creatinine, inclusive at Screening).
8. Has glycosylated hemoglobin (HbA1c) less than or equal to 10.5% at screening.
9. If a subject is regularly using dipeptidyl peptidase-4 inhibitor (DPP-4i) or sodium-glucose cotransporter 2 inhibitor (SGLT2i) to treat diabetes, he/she has been on a stable dose and regimen within 2 months prior to Screening.
10. All participants who are not surgically sterile or post-menopausal, or whose partners are not surgically-sterile or postmenopausal, must use two effective birth control methods or abstain from intercourse during this study.

Exclusion Criteria:

1. Has received any investigational compound within 90 days prior to Screening.
2. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
3. Is taking any combination of dual renin-angiotensin system (RAS) inhibition (such as an ACE inhibitor and an ARB or an ACE inhibitor and a mineralocorticoid receptor antagonist).
4. Has type 1 diabetes mellitus or a history of ketoacidosis.
5. Has poorly-controlled blood pressure (systolic blood pressure >160 or diastolic blood pressure >110, with blood pressure measured in the seated position after at least 5 minutes of rest) at Screening and Day 1.
6. Has received dialysis within 3 months of Screening.
7. Has infectious diseases or leg ulcers at Screening (all per discretion of Principal Investigator [PI]).
8. Has severe concurrent disease which, in the judgment of the investigator, would interfere significantly with the assessments of safety and efficacy during this study.
9. Has known infection with human immunodeficiency virus (HIV), or a positive test for Hepatitis B, Hepatitis C, or tuberculosis (TB) at Screening. Subjects who have a positive TB skin test at Screening must rule out active or latent tuberculosis documented by chest x-ray in order to be considered eligible for study participation.
10. Has used long-term immune suppressants, steroid therapy (except for topical use or inhalation), chronic use of non-steroidal anti-inflammatory drug (NSAIDs), cyclooxygenase type 2 (COX-2) inhibitors within 2 weeks prior to Screening. Short-term use is defined as a duration of ≤4 weeks of continuous use.
11. In the judgment of the principal investigator, participants who are likely to be non-compliant or uncooperative during the study.
12. Has known non-diabetic kidney disease (such as autosomal dominant polycystic kidney disease (ADPCKD), Immunoglobulin A (IgA) nephropathy, focal segmental glomerulosclerosis, or obstructive uropathy). Hypertensive nephrosclerosis superimposed on diabetic kidney disease is acceptable.
13. Had a previous renal transplant.
14. Has hypersensitivity to other monoclonal antibodies (mAb) or to any component of the formulation of MLN1202.
15. Has history of malignancy within the previous 5 years (with the exception of adequately treated basal cell or squamous cell carcinoma of the skin).
16. Is symptomatic with dysuria, and has a positive urine culture at screening.
17. If female, the subject is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period and for 56 days (8weeks) afterwards.
18. If male, the subject intends to donate sperm during the course of this study or for 12 weeks thereafter.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2015-11-17 (Actual); Study Completion 2015-11-17 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Urinary Albumin-to-Creatinine Ratio (UACR) at Day 85 | Baseline and Day 85
  UACR will be calculated using the geometric mean of 3 consecutive days first in the morning urine voids. First morning void is defined as a void upon awakening and before beginning daily activities.

SECONDARY OUTCOMES:
Change from Baseline in Urinary Albumin-to-Creatinine Ratio (UACR) Over Time | Baseline and Days 29, 57, 85, and 113
  For Days 29 and 57 UACR will be evaluated from a single first morning void. For Days 85 and 113 UACR will be calculated using the geometric mean of 3 consecutive days first in the morning urine voids. First morning void is defined as a void upon awakening and before beginning daily activities.
Change from Baseline in Urinary Protein:Creatinine Ratio (UPCR) Over Time | Baseline and Days 29, 57, 85, and 113
  For Days 29 and 57 UPAR will be evaluated from a single first morning void. For Days 85 and 113 UPCR will be calculated using the geometric mean of 3 consecutive days first in the morning urine voids. First morning void is defined as a void upon awakening and before beginning daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda